CLINICAL TRIAL: NCT01007253
Title: Effect of Veramyst and Olopatadine 0.2% Opthalmic Solution Alone and In Combination on the Nasal and Ocular Symptoms of the Early Reaction to Nasal Challenge With Allergen.
Brief Title: Effect of Veramyst and Olopatadine 0.2% Opthalmic Solution on Allergy Symptoms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Robert Naclerio, MD, University of Chicago
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 09-287-B
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Results first posted 2013-07-17 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-06

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — fluticasone furoate; Fluticasone; Olopatadine Hydrochloride; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- FF/PL, PL/OLO, FF/OLO, PL/PL (Other): Each subject received a total of 4 weeks of treatment (1 week per treatment with 2 week washout period between treatments) in the following order:
  * fluticasone furoate (FF) nasal spray and PL eye drops (FF/PL)
  * PL nasal spray and olopatadine (OLO) 0.2% ophthalmic solution (PL/OLO),
  * FF nasal spray and olopatadine (OLO) 0.2% ophthalmic solution (FF/OLO), and
  * placebo (PL) nasal spray and PL eye drops (PL/PL).
  Interventions: Drug: PL nasal spray; Drug: fluticasone furoate (FF); Drug: PL eye drops; Drug: olopatadine (OLO)
- PL/OLO, FF/OLO, PL/PL, FF/PL (Other): Each subject received a total of 4 weeks of treatment (1 week per treatment with 2 week washout period between treatments) in the following order:
  * PL nasal spray and olopatadine (OLO) 0.2% ophthalmic solution (PL/OLO),
  * FF nasal spray and olopatadine (OLO) 0.2% ophthalmic solution (FF/OLO),
  * placebo (PL) nasal spray and PL eye drops (PL/PL), and
  * fluticasone furoate (FF) nasal spray and PL eye drops (FF/PL).
  Interventions: Drug: PL nasal spray; Drug: fluticasone furoate (FF); Drug: PL eye drops; Drug: olopatadine (OLO)
- FF/OLO, PL/PL, FF/PL, PL/OLO (Other): Each subject received a total of 4 weeks of treatment (1 week per treatment with 2 week washout period between treatments) in the following order:
  * FF nasal spray and olopatadine (OLO) 0.2% ophthalmic solution (FF/OLO),
  * placebo (PL) nasal spray and PL eye drops (PL/PL),
  * fluticasone furoate (FF) nasal spray and PL eye drops (FF/PL), and
  * PL nasal spray and olopatadine (OLO) 0.2% ophthalmic solution (PL/OLO).
  Interventions: Drug: PL nasal spray; Drug: fluticasone furoate (FF); Drug: PL eye drops; Drug: olopatadine (OLO)
- PL/PL, FF/PL, PL/OLO, FF/OLO (Other): Each subject received a total of 4 weeks of treatment (1 week per treatment with 2 week washout period between treatments) in the following order:
  * placebo (PL) nasal spray and PL eye drops (PL/PL),
  * fluticasone furoate (FF) nasal spray and PL eye drops (FF/PL),
  * PL nasal spray and olopatadine (OLO) 0.2% ophthalmic solution (PL/OLO), and
  * FF nasal spray and olopatadine (OLO) 0.2% ophthalmic solution (FF/OLO).
  Interventions: Drug: PL nasal spray; Drug: fluticasone furoate (FF); Drug: PL eye drops; Drug: olopatadine (OLO)

INTERVENTIONS:
Drug: PL nasal spray — 2 puffs of PL nasal spray (from GlaxoSmithKline) in each nostril once a day for 1 week
Drug: fluticasone furoate (FF) — 2 puffs of FF nasal spray in each nostril once a day for 1 week
  Other Names: Veramyst
Drug: PL eye drops — 1 drop of placebo eye drops (lubricant eye drops with active ingredients 0.3% glycerin) in each eye once a day for 1 week
Drug: olopatadine (OLO) — 1 drop of OLO eye drops in each eye once a day for 1 week
  Other Names: Olopatadine 0.2% ophthalmic solution

SUMMARY:
People who have hayfever or allergic rhinitis often complain about eye symptoms associated with their nasal symptoms. How people with hayfever develop eye symptoms is not clear. The purpose of this study is to better understand the generation of eye symptoms in patients with allergic rhinitis. We have previously shown that placing the substance that subjects are allergic to in their nose causes both nose and eye symptoms. This can be explain by a parasympathetic neurogenic reflex from the nose to the eye. Such a reflex would readily explain the tearing and watery eye symptoms, but does not explain the itch. In this study, we are going to address one possible explanation for the itch; does an axonal neurogenic reflex stimulate mast cells in the eye to release histamine, which then causes the itch? We will do this by placing an antihistamine drop in the eye and challenge the nose with allergen. We will also attempt to demonstrate that mast activation isn't effected by blocking the initiating of the reflex with a nasal steroid, as done in our previous study, and showing that the addition of an antihistamine does not add to the reduction of symptoms.

DETAILED DESCRIPTION:
We performed a randomized, double-blind, double-dummy, placebo-controlled, four-way crossover study in 21 subjects with seasonal allergic rhinitis studied out of season. Healthy patients, between 18 and 50 years of age, came to the Nasal Physiology Laboratory at The University of Chicago for screening, where they completed an allergy questionnaire and underwent skin puncture testing for confirmation of allergy to grass or ragweed. Female subjects were given pregnancy tests. Patients who were eligible then underwent a screening nasal challenge with either grass or ragweed allergen depending on their skin test results and history. The study was approved by the Institutional Review Board at The University of Chicago and all of the patients gave written informed consent before entry.

After a 2-week washout period, after the screening challenge, 21 subjects who had positive screening challenge returned to the Nasal Physiology Laboratory where they were randomized to receive 1 week of one of four treatments:

* placebo (PL) nasal spray and PL eye drops (PL/PL),
* PL nasal spray and olopatadine (OLO) 0.2% ophthalmic solution (PL/OLO),
* fluticasone furoate (FF, also known as Veramyst) nasal spray and PL eye drops (FF/PL), and
* FF nasal spray and olopatadine (OLO) 0.2% ophthalmic solution (FF/OLO).

Specifically, the PL eye drops used were lubricant eye drops with active ingredients of 0.3% glycerin and 1.0% propylene glycol and the PL nasal spray was provided by GlaxoSmithKline. Treatment with OLO consisted of 1 drop of 0.2% OLO in each eye daily and treatment of FF consisted of 2 puffs in each nostril daily, giving a total of 110 micrograms delivered in each nostril. After a week of each of the treatments, the subjects returned to the Nasal Physiology Laboratory to undergo a nasal challenge. The subjects then returned the next day while still receiving treatment for another nasal challenge to augment the nasal ocular reflex. Next, the patients had a 2-week washout period and then switched over to the next randomized treatment arm. This sequence was repeated until subjects completed all four arms of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18 and 45 years of age.
2. History of grass and/or ragweed allergic rhinitis.
3. Positive skin test to grass and/or ragweed antigen.
4. Positive response to screening nasal challenge.

Exclusion Criteria:

1. Physical signs or symptoms suggestive of renal, hepatic or cardiovascular disease.
2. Pregnant or lactating women.
3. Upper respiratory infection within 14 days of study start.
4. forced expiratory volume at one second (FEV1) <80% of predicted at screening for subjects with history of mild asthma.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2009-11; Primary Completion 2010-04 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Naclerio, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Result] Baroody FM, Logothetis H, Vishwanath S, Bashir M, Detineo M, Naclerio RM. Effect of intranasal fluticasone furoate and intraocular olopatadine on nasal and ocular allergen-induced symptoms. Am J Rhinol Allergy. 2013 Jan;27(1):48-53. doi: 10.2500/ajra.2013.27.3841. PMID 23406601

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy patients age 18-50 completed an allergy questionnaire and underwent skin puncture testing for confirmation of allergy to grass or ragweed. Female subjects were given pregnancy tests. Patients who were eligible then underwent a screening nasal challenge with either grass or ragweed allergen depending on their skin test results and history.
Pre-assignment Details: After a 2-week washout period, 21 subjects who had positive screening challenge returned to the Nasal Physiology Laboratory where they were randomized to receive one of four treatment orderings in this four-way crossover study.
Period: First Intervention
Arm/Group | FF/PL, PL/OLO, FF/OLO, PL/PL | PL/OLO, FF/OLO, PL/PL, FF/PL | FF/OLO, PL/PL, FF/PL, PL/OLO | PL/PL, FF/PL, PL/OLO, FF/OLO
Started | 6 | 5 | 5 | 5
Completed | 6 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period (2 Weeks) # 1
Arm/Group | FF/PL, PL/OLO, FF/OLO, PL/PL | PL/OLO, FF/OLO, PL/PL, FF/PL | FF/OLO, PL/PL, FF/PL, PL/OLO | PL/PL, FF/PL, PL/OLO, FF/OLO
Started | 6 | 5 | 5 | 5
Completed | 6 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | FF/PL, PL/OLO, FF/OLO, PL/PL | PL/OLO, FF/OLO, PL/PL, FF/PL | FF/OLO, PL/PL, FF/PL, PL/OLO | PL/PL, FF/PL, PL/OLO, FF/OLO
Started | 6 | 5 | 5 | 5
Completed | 6 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period (2 Weeks) # 2
Arm/Group | FF/PL, PL/OLO, FF/OLO, PL/PL | PL/OLO, FF/OLO, PL/PL, FF/PL | FF/OLO, PL/PL, FF/PL, PL/OLO | PL/PL, FF/PL, PL/OLO, FF/OLO
Started | 6 | 5 | 5 | 5
Completed | 6 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Third Intervention
Arm/Group | FF/PL, PL/OLO, FF/OLO, PL/PL | PL/OLO, FF/OLO, PL/PL, FF/PL | FF/OLO, PL/PL, FF/PL, PL/OLO | PL/PL, FF/PL, PL/OLO, FF/OLO
Started | 6 | 5 | 5 | 5
Completed | 6 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period (2 Weeks) # 3
Arm/Group | FF/PL, PL/OLO, FF/OLO, PL/PL | PL/OLO, FF/OLO, PL/PL, FF/PL | FF/OLO, PL/PL, FF/PL, PL/OLO | PL/PL, FF/PL, PL/OLO, FF/OLO
Started | 6 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5
Not Completed | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Period: Fourth Intervention
Arm/Group | FF/PL, PL/OLO, FF/OLO, PL/PL | PL/OLO, FF/OLO, PL/PL, FF/PL | FF/OLO, PL/PL, FF/PL, PL/OLO | PL/PL, FF/PL, PL/OLO, FF/OLO
Started | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive PL/PL first, FF/PL first, PL/OLO first, and FF/OLO first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 21
Age Continuous [Mean (Standard Deviation); unit: years] | 31.1 (6.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Total Eye Symptoms Score Difference
Description: After treatment, each participant was subjected to a diluent (control) challenge in one eye and was asked to rate 2 eye symptoms (watery and itchy) according to the following scale: 0=none, 1=mild, 2=moderate, 3=severe. The participant was then exposed to 3 doses of an antigen challenge and was asked to similarly rate severity of watery and itchy eye symptoms after each dose. Diluent challenge scores were subtracted from the scores recorded after each dose. This process was repeated in the other eye. The outcome is the total of the score differences (i.e. score after each dose subtracted by diluent challenge score) summed across doses, symptoms (watery and itchy), and eyes (left and right). Thus, each participant's total score is an integer value ranging from -36 to 36.
Time Frame: 50 minutes [duration of 3 nasal challenges and 2 washout periods]
Population: One subject was removed from the study due to upper respiratory tract infection, reducing the number of evaluable subjects from 21 to 20.
Measure: Median (Full Range); unit: units on a scale
Groups:
- PL/PL: placebo (PL) nasal spray and PL eye drops
- FF/PL: fluticasone furoate (FF) nasal spray and PL eye drops
- PL/OLO: PL nasal spray and olopatadine (OLO) 0.2% ophthalmic solution
- FF/OLO: FF nasal spray and olopatadine (OLO) 0.2% ophthalmic solution
Arm/Group | PL/PL | FF/PL | PL/OLO | FF/OLO
Number analyzed (Participants) | 20 | 20 | 20 | 20
units on a scale | 6 [0 to 23] | 0 [-6 to 11] | 2.5 [0 to 26] | 1.5 [-9 to 16]
Statistical Analysis 1: Comparison: PL/PL vs FF/PL vs PL/OLO vs FF/OLO; Analysis of variance (ANOVA) was used to test the null hypothesis of no mean eye symptoms score difference among the four treatment groups; Test type: Superiority or Other; p < 0.001, Friedman ANOVA

2. Secondary Outcome: Total Nasal Symptoms Score Difference
Description: After treatment, each participant was subjected to a diluent (control) challenge in one nostril and was asked to rate nasal symptoms (congestion, rhinorrhea, and itchy nose/throat) according to the following scale: 0=none, 1=mild, 2=moderate, 3=severe. The participant was then exposed to 3 doses of an antigen challenge and was asked to similarly rate severity of nasal symptoms after each dose. Diluent challenge scores were subtracted from the scores recorded after each dose. This process was repeated in the other nostril. The outcome is the total number of score differences (i.e. score after each dose subtracted by diluent challenge score) summed across doses, symptoms (congestion, rhinorrhea, and itchy nose/throat), and nostrils (left and right). Thus, each participant's total score is an integer value ranging from -36 to 36.
Time Frame: 50 minutes [duration of 3 nasal challenges and 2 washout periods]
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | PL/PL | FF/PL | PL/OLO | FF/OLO
Number analyzed (Participants) | 20 | 20 | 20 | 20
units on a scale | 17 [6 to 34] | 10 [3 to 31] | 9 [-2 to 35] | 9 [0 to 26]
Statistical Analysis 1: Comparison: PL/PL vs FF/PL vs PL/OLO vs FF/OLO; Analysis of variance (ANOVA) was used to test the null hypothesis of no mean nasal symptoms score difference among the four treatment groups; Test type: Superiority or Other; p = 0.05, Friedman ANOVA

3. Secondary Outcome: Total Number of Sneezes
Time Frame: 50 minutes [duration of 3 nasal challenges and 2 washout periods]
Population: as for outcome 1
Measure: Median (Full Range); unit: sneezes
Arm/Group | PL/PL | FF/PL | PL/OLO | FF/OLO
Number analyzed (Participants) | 20 | 20 | 20 | 20
sneezes | 10 [0 to 36] | 2.5 [0 to 50] | 2.5 [0 to 49] | 1.0 [0 to 16]
Statistical Analysis 1: Comparison: PL/PL vs FF/PL vs PL/OLO vs FF/OLO; Analysis of variance (ANOVA) was used to test the null hypothesis of no mean sneeze difference among the four treatment groups; Test type: Superiority or Other; p = 0.001, Friedman ANOVA

4. Secondary Outcome: Change in Histamine Level (Across Nasal Challenges)
Description: Histamines are simple chemical substances produced by immune system cells when reacting to an antigen in response to foreign invaders like germs and bacteria.
  Histamine in nasal lavages was measured using a histamine enzyme immunoassay kit market by SPI-BIo, Bertin Pharma (Montigny le Bretonneux, France). The limit of detection of the assay is 0.4 nM, and levels below the detection limit were arbitrarily assigned a value of 0.2 nM. Samples that yielded values above the upper detection limit of the assay were diluted and reassayed.
  For each patient, histamine levels recorded after the diluent challenge were subtracted from histamine levels recorded after each of the three nasal challenges. These differences were added across challenges, yielding the total change in histamine level reported in this outcome for each patient.
Time Frame: 50 minutes [duration of 3 nasal challenges and 2 washout periods]
Population: as for outcome 1
Measure: Median (Full Range); unit: nM
Arm/Group | PL/PL | FF/PL | PL/OLO | FF/OLO
Number analyzed (Participants) | 20 | 20 | 20 | 20
nM | 5.9 [-2 to 203] | 0.3 [-91 to 209] | 11.4 [-9 to 435] | 3.4 [-34 to 250]
Statistical Analysis 1: Comparison: PL/PL vs FF/PL vs PL/OLO vs FF/OLO; Analysis of variance (ANOVA) was used to test the null hypothesis of no mean histamine level difference among the four treatment groups; Test type: Superiority or Other; p = 0.11, Friedman ANOVA

5. Secondary Outcome: Change in Tryptase Level (Across Nasal Challenges)
Description: Tryptase is an enzyme that is released, along with histamine and other chemicals, from mast cells when they are activated, often as part of an allergic immune response. Tryptase in nasal lavages was measured using the ImmunoCap tryptase assay, by Phadia (Uppsala, Sweden). The limit of detection of the assay is 1.0 ng/mL, and levels below this value were arbitrarily assigned a value of 0.5 ng/mL.
  For each patient, tryptase levels recorded after the diluent challenge were subtracted from tryptase levels recorded after each of the three nasal challenges. These differences were added across challenges, yielding the total change in tryptase level reported in this outcome for each patient.
Time Frame: 50 minutes [duration of 3 nasal challenges and 2 washout periods]
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/mL
Arm/Group | PL/PL | FF/PL | PL/OLO | FF/OLO
Number analyzed (Participants) | 20 | 20 | 20 | 20
ng/mL | 5 [0 to 527] | 0 [0 to 21] | 2 [0 to 140] | 0 [0 to 49]
Statistical Analysis 1: Comparison: PL/PL vs FF/PL vs PL/OLO vs FF/OLO; Analysis of variance (ANOVA) was used to test the null hypothesis of no mean tryptase level difference among the four treatment groups; Test type: Superiority or Other; p < 0.001, Friedman ANOVA

6. Secondary Outcome: Total Number of Eosinophils
Description: The percentage of eosinophils among white blood cells was determined under light microscopy at 1000x magnification, and the total number of eosinophils in each lavage was then calculated. The specimens that had no eosinophils identified on differential counting despite adequate cells on the smear were assigned a number that corresponded to the lowest number of eosinophils on a slide where the number could be counted. That number was 33 total eosinophils.
Time Frame: 50 minutes [duration of 3 nasal challenges and 2 washout periods]
Population: as for outcome 1
Measure: Median (Full Range); unit: eosinophils
Arm/Group | PL/PL | FF/PL | PL/OLO | FF/OLO
Number analyzed (Participants) | 20 | 20 | 20 | 20
eosinophils | 7883 [33 to 2246440] | 238 [33 to 604800] | 9606 [33 to 953250] | 311 [33 to 224000]

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | PL/PL | FF/PL | PL/OLO | FF/OLO
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/21 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes